CLINICAL TRIAL: NCT00616629
Title: A Multi-centre, Double-blind, Randomised, Placebo-controlled, Singledose, Phase II Study to Assess the Effects on Atrial and Ventricular Refractoriness and Haemodynamics of an Intravenous Infusion of AZD1305 in Patients Undergoing an Invasive Electrophysiological Procedure
Brief Title: Cardiac Electrophysiological Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca AZD1305 Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D3190C00005; 2007-0003455-36 (EudraCT No)
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-08

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter | interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD1305 — Intravenous infusion

SUMMARY:
The purpose of the study is to measure the effects of AZD1305 on cardiac electrophysiological properties and intracardiac pressures

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial flutter (with a ventricular rate of <100 beats/minute at enrolment), scheduled for curative catheter ablation
* Sinus rhythm at randomisation

Exclusion Criteria:

* QTc (Fridericia, QTcF ) >450 ms measured in sinus rhythm at randomisation,
* Serum potassium below 3.8 or above 5.0 mmol/L or plasma potassium below 3.6 or above 5.0 mmol/L
* QRS duration >120 ms at randomisation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Toivonen, MD, Principal Investigator — Helsinki University Central Hospital
Locations (13):
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Copenhagen
  - Research Site, Hellerup
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Oulu
- Norway (2):
  - Research Site, Bergen
  - Research Site, Oslo
- Sweden (4):
  - Research Site, Gŏteborg
  - Research Site, Linkŏping
  - Research Site, Ŏrebro
  - Research Site, Umeå

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 68 patients were enrolled into the study. The study randomised 55 patients and 50 of those patients received study drug. All patients who received study drug completed the study.
Pre-assignment Details: At the pre-entry visit, which took place within 14 days before the planned catheter ablation (Study Day), patients underwent a full clinical assessment including a physical examination, ECG recording, Bood pressure(BP)/heart rate measurement, routine laboratory tests, and transthoracic echocardiography (TTE, if not done within the prior 6 months).
Groups:
- AZD1305 Dose Group 1: Loading dose 15 min at 43.5 mg/h, Maintenance dose maximum 60 additional min at 19.6 mg/h
- AZD1305 Dose Group 2: Loading dose 15 min at 130.4 mg/h, Maintenance dose maximum 60 additional min at 58.7 mg/h
- AZD1305 Dose Group 3: Loading dose 15 min at 325.9 mg/h, Maintenance dose maximum 60 additional min at 146.6 mg/h
- AZD1305 Dose Group 4: Loading dose 15 min at 488.8 mg/h, Maintenance dose maximum 60 additional min at 220.0 mg/h
- Placebo: Corresponding placebo
Period: Overall Study
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Started | 13 (Two patients never received study drug) | 14 (Two patients never received study drug) | 14 (One patient never received study drug) | 2 | 12
Completed | 11 | 12 | 13 | 2 | 12
Not Completed | 2 | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 1 | 0 | 0
Not completed — AV-block | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 13 | 2 | 12 | 50
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age (years) | 60 (14) | 62 (6) | 60 (8) | 50 (23) | 62 (6) | 56 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 0 | 0 | 6
  Male | 9 | 10 | 11 | 2 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: LAERP (Left Atrial Effective Refractory Period (ie, the Longest S1-S2 Interval That Fails to Result in Atrial Depolarisation))
Description: Absolute change, after - before infusion
Time Frame: Measurements were obtained twice, from the invasive electrophysiological measurements made before and 20 min (or more) after the start of administration of the investigational product
Measure: Mean (Full Range); unit: ms
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 11 | 11 | 13 | 2 | 11
ms | 11 (-15) [-15 to 40] | 43 (0) [0 to 210] | 55 (-5) [-5 to 85] | 50 (40) [40 to 60] | -10 (-90) [-90 to 30]

2. Secondary Outcome: RAERP (Right Atrial Effective Refractory Period)
Description: Absolute change, after - before infusion
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: ms
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 11 | 12 | 12 | 2 | 11
ms | 19 (-5) [-5 to 40] | 42 (0) [0 to 75] | 84 (-30) [-30 to 165] | 135 (100) [100 to 170] | -12 (-90) [-90 to 40]

3. Secondary Outcome: VERP (Ventricular Effective Refractory Period)) and Other Electrophysiological and Electrocardiographic Variables; RR, P Wave Duration, PR, QRS, QTend, QTcF, QTtop, QTend - QTtop)
Description: Absolute change, after - before infusion
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: ms
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 2 | 11
ms | 11 (-25) [-25 to 30] | 41 (5) [5 to 145] | 59 (25) [25 to 110] | 65 (45) [45 to 85] | 3 (-25) [-25 to 40]

4. Secondary Outcome: QTcF (Interval From the Beginning of the Q or R Wave to the End of the T Wave in the Surface ECG, Corrected for Changes in RR Interval Using Fridericia' Formula =QT/RR1/3 Interval in Seconds)
Description: Absolute change, after - before infusion
Time Frame: Measurements were obtained twice, from the invasive electrophysiological measurements made before and 20 min (or more) after the start of administration of the investigational product. ECG measurements, including QTcF, are available from several additiona
Measure: Mean (Full Range); unit: ms
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 2 | 12
ms | 20 (-2) [-2 to 42] | 65 (13) [13 to 150] | 79 (31) [31 to 128] | 65 (59) [59 to 70] | 4 (-51) [-51 to 47]

5. Secondary Outcome: Cmax Observed for AZD1305
Description: A total of 13 scheduled PK samples for each patient during and after infusion
Time Frame: During and after infusion
Measure: Mean (Full Range); unit: umol/L
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 2 | 0
umol/L | 0.178 (0.104) [0.104 to 0.279] | 0.692 (0.368) [0.368 to 1.82] | 1.46 (0.931) [0.931 to 2.81] | 2.41 (2.24) [2.24 to 2.58] |

6. Secondary Outcome: AUC Total of AZD1305 (Umol*h/L)
Description: A total of 13 scheduled PK samples for each patient during and after infusion
Time Frame: Based on PK samples during and after infusion
Measure: Mean (Full Range); unit: umol*h/L
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 2 | 0
umol*h/L | 1.54 (0.97) [0.97 to 2.21] | 4.97 (2.70) [2.70 to 10.0] | 10.3 (5.71) [5.71 to 18.9] | 17.3 (16.5) [16.5 to 18.2] |

7. Secondary Outcome: Number of Patients Who Had at Least One AE
Description: Number of patients
Time Frame: During active treatment period
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Number analyzed (Participants) | 11 | 12 | 13 | 2 | 12
Participants | 2 | 2 | 2 | 1 | 1

ADVERSE EVENTS:
Arm/Group | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/12 | 1/13 | 0/2 | 1/12
Other Adverse Events (participants affected / at risk) | 2 | 1 | 1 | 1 | 0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1305 Dose Group 1 (N=11) | AZD1305 Dose Group 2 (N=12) | AZD1305 Dose Group 3 (N=13) | AZD1305 Dose Group 4 (N=2) | Placebo (N=12)
Bradycardia And Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AZD1305 Dose Group 1 | AZD1305 Dose Group 2 | AZD1305 Dose Group 3 | AZD1305 Dose Group 4 | Placebo
Atrial Fibrillation (Cardiac disorders) | 1/11 | 0/12 | 0/13 | 0/2 | 0/12
Muscoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1/11 | 0/12 | 0/13 | 0/2 | 0/12
Vision Blurred (Eye disorders) | 0/11 | 1/12 | 0/13 | 0/2 | 0/12
Syncope Vasovagal (Nervous system disorders) | 0/11 | 0/12 | 1/13 | 0/2 | 0/12
Vomiting (Gastrointestinal disorders) | 0/11 | 0/12 | 0/13 | 1/2 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less